CLINICAL TRIAL: NCT03733301
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Combination With Topical Corticosteroids in Adult Patients With Moderate to Severe Atopic Dermatitis BREEZE-AD7
Brief Title: A Study of Baricitinib (LY3009104) in Combination With Topical Corticosteroids in Adults With Moderate to Severe Atopic Dermatitis
Acronym: BREEZE-AD7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17100; I4V-MC-JAIY (Other: Eli Lilly and Company); 2018-001726-26 (EudraCT Number)
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4 Milligram (mg) Baricitinib (Experimental): 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids (TCS). Placebo administered orally once daily to match 2 mg Baricitinib.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid; Drug: Placebo
- 2 mg Baricitinib (Experimental): 2 mg Baricitinib administered orally once daily in combination with TCS. Placebo administered orally once daily to match 4 mg Baricitinib.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid; Drug: Placebo
- Placebo (Placebo Comparator): Placebo administered orally once daily in combination with TCS.
  Interventions: Drug: Topical corticosteroid; Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 2 mg Baricitinib; 4 Milligram (mg) Baricitinib
Drug: Topical corticosteroid — Administered as standard-of-care.
Drug: Placebo — Administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of baricitinib in combination with topical corticosteroids (TCS) in participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with moderate to severe atopic dermatitis for at least 12 months.
* Have had inadequate response to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episodes of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to randomization.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor less than 4 weeks prior to randomization.
  * Received any parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
  * Have had an intra-articular corticosteroid injection within 6 weeks prior to planned randomization.
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (68):
- Argentina (5):
  - Centro de Investigaciones Metabólicas (CINME) - Comite, Ciudad Autonoma Buenos Aires
  - Fundacion CIDEA, Ciudad Autonoma Buenos Aires
  - Instituto de Neumonología y Dermatología, Ciudad Autonoma Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, Ciudad Autonoma Buenos Aires
  - Parra Dermatología, Mendoza
- Australia (7):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Clinical Trials SA Pty Ltd, Adelaide, South Australia
  - Skin and Cancer Foundation Inc., Melbourne, Victoria
  - Fremantle Dermatology, Perth, Western Australia
- Universitätsklinikum Graz, Graz, Styria, Austria
- Germany (10):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Rosenpark Research Geschäftsbereich der Rosenparkklinik GmbH, Darmstadt, Hesse
  - Dermatologisches Zentrum Osnabrück Nord, Bramsche, Lower Saxony
  - Universitätsklinikum Aachen - UKA, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Berlin
  - TFS Trial Form Support GmbH, Hamburg
- Italy (5):
  - Policlinico Univ. Agostino Gemelli, Rome, Lazio
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Ospedale San Martino di Genova, Genova
  - Azienda Ospedaliera - Universitaria Pisana, Pisa
  - ULSS 8 UOC Dermatologia Viale Rodolfi, 37, Vicenza
- Japan (17):
  - Kawashima Dermatology Clinic, Ichikawa-shi, Chiba
  - Medical Corporation Soleil Miyata Dermatology Clinic, Matsudo-shi, Chiba
  - Yamano Dermatological Clinic, Dazaifu, Fukuoka
  - Tashiro Dermatological Clinic, Iizuka, Fukuoka
  - Shibaki Dermatology Clinic, Sapporo, Hokkaido
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Queen's Square Dermatology and Allergology, Nishi-ku, Yokohama-city, Kanagawa
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Senri-Chuo Hanafusa Dermatology Clinic, Toyonaka-shi, Osaka
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Iidabashi Clinic, Chiyoda-ku, Tokyo
  - Tokyo Teishin Hospital, Chiyoda-Ku, Tokyo
  - Hosono Clinic, Chuo-ku, Tokyo
  - Oizumi Hanawa Clinic, Nerima-ku, Tokyo
  - Yamate Dermatological Clinic, Shinjuku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - Shirasaki Clinic, Takaoka-shi, Toyama
- Poland (4):
  - Dermed Centrum Medyczne Sp. z o.o., Lodz
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Centrum Medyczne AMED, Warsaw
  - Centrum Medyczne Evimed, Warsaw
- South Korea (8):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Korea
  - Severance Hospital Yonsei University Health System, Seoul
  - Konkuk University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Chungang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
- Taiwan (6):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Taipei, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan, (r.o.c.)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Wollenberg A, Kircik L, Simpson E, Brinker D, Katoh N, Rueda MJ, Issa M, Yang F, Feely M, Alexis A. Pooled Analysis of Baricitinib Tolerability in Patients With Atopic Dermatitis in Relation to Acne, Headache, and Gastrointestinal Events From 8 Clinical Trials. Dermatitis. 2023 Jul-Aug;34(4):308-314. doi: 10.1089/derm.2022.0027. Epub 2023 Feb 6. PMID 36749121
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] Thyssen JP, Buhl T, Fernandez-Penas P, Kabashima K, Chen S, Lu N, DeLozier AM, Casillas M, Stander S. Baricitinib Rapidly Improves Skin Pain Resulting in Improved Quality of Life for Patients with Atopic Dermatitis: Analyses from BREEZE-AD1, 2, and 7. Dermatol Ther (Heidelb). 2021 Oct;11(5):1599-1611. doi: 10.1007/s13555-021-00577-x. Epub 2021 Jul 18. PMID 34275122
- [Derived] Buhl T, Rosmarin D, Serra-Baldrich E, Fernandez-Penas P, Igarashi A, Konstantinou MP, Chen S, Lu N, Pierce E, Casillas M. Itch and Sleep Improvements with Baricitinib in Patients with Atopic Dermatitis: A Post Hoc Analysis of 3 Phase 3 Studies. Dermatol Ther (Heidelb). 2021 Jun;11(3):971-982. doi: 10.1007/s13555-021-00534-8. Epub 2021 Apr 25. PMID 33899152
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- [Derived] Reich K, Kabashima K, Peris K, Silverberg JI, Eichenfield LF, Bieber T, Kaszuba A, Kolodsick J, Yang FE, Gamalo M, Brinker DR, DeLozier AM, Janes JM, Nunes FP, Thyssen JP, Simpson EL. Efficacy and Safety of Baricitinib Combined With Topical Corticosteroids for Treatment of Moderate to Severe Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2020 Dec 1;156(12):1333-1343. doi: 10.1001/jamadermatol.2020.3260. PMID 33001140
- See also: A Study of Baricitinib (LY3009104) in Combination With Topical Corticosteroids in Adults With Moderate to Severe Atopic Dermatitis — https://www.lillytrialguide.com/en-US/studies/atopic-dermatitis/JAIY

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 16-week treatment period had an option to enter extension study JAHN (NCT03334435).
Groups:
- Placebo: Placebo administered orally once daily.
- 2 mg Baricitinib: 2 mg Baricitinib administered orally once daily.
- 4 mg Baricitinib: 4 mg Baricitinib administered orally once daily.
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Started | 109 | 109 | 111
Received One Dose of Study Drug | 108 | 109 | 111
Completed | 102 | 100 | 107
Not Completed | 7 | 9 | 4
Not completed — Screen Fail | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Total
Number analyzed (Participants) | 109 | 109 | 111 | 329
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 106 | 105 | 111 | 322
  >=65 years | 3 | 4 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 36 | 113
  Male | 71 | 70 | 75 | 216
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 57 | 57 | 54 | 168
  Multiple | 6 | 2 | 3 | 11
  White | 46 | 50 | 54 | 150
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 8 | 6 | 11 | 25
  South Korea | 29 | 19 | 15 | 63
  Austria | 2 | 1 | 5 | 8
  Japan | 21 | 20 | 22 | 63
  Taiwan | 9 | 12 | 15 | 36
  Poland | 11 | 9 | 6 | 26
  Italy | 7 | 6 | 6 | 19
  Australia | 4 | 14 | 9 | 27
  Germany | 12 | 18 | 17 | 47
  Spain | 6 | 4 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement
Description: The IGA measures investigators global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 14.7 | 23.9 | 30.6
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.082, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.92 to 3.85]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.38 to 5.56]

2. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 22.9 | 43.1 | 47.7
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.44 to 4.76]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.80 to 5.97]

3. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 13.8 | 16.5 | 24.3
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.574, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.59 to 2.62]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.045, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.02 to 4.20]

4. Secondary Outcome: Percent Change From Baseline on EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Squares Mean (LSM) were calculated using mixed model repeated measures (MMRM) with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit interaction as fixed categorical effects and baseline score and baseline score-by-visit interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants who had Week 16 EASI data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 90 | 100 | 100
percent change | -45.08 (3.828) | -58.16 (3.689) | -67.21 (3.679)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -13.08, 95% CI 2-sided [-23.42 to -2.73], Standard Error of Mean 5.256
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -22.13, 95% CI 2-sided [-32.48 to -11.78], Standard Error of Mean 5.259

5. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 7.3 | 11.0 | 18.0
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.364, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.61 to 3.81]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.15 to 6.34]

6. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 16
Population: All randomized participants with Baseline Itch Score >= 4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 104 | 97 | 100
percentage of participants | 20.2 | 38.1 | 44.0
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.48 to 5.61]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.84, 95% CI 2-sided [1.98 to 7.46]

7. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS)
Description: The ADSS is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep due to itch, frequency of waking due to itch, and difficulty getting back to sleep last night due to itch. Item 2 frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times, where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually. LS Mean were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit interaction as fixed categorical effects and baseline score and baseline score-by-visit interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 ADSS Item 2 (frequency of waking) data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 98 | 94
units on a scale | -0.51 (0.151) | -1.33 (0.147) | -1.42 (0.147)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.23 to -0.41], Standard Error of Mean 0.209
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.33 to -0.51], Standard Error of Mean 0.209

8. Secondary Outcome: Change From Baseline in Skin Pain NRS
Description: Skin Pain NRS is a patient-administered,11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours. LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Skin Pain NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 2 mg Baricitinib: Baricitinib 2 mg administered orally once daily.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 98 | 94
units on a scale | -2.06 (0.231) | -3.22 (0.224) | -3.73 (0.226)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.78 to -0.52], Standard Error of Mean 0.319
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.66, 95% CI 2-sided [-2.30 to -1.30], Standard Error of Mean 0.322

9. Secondary Outcome: Percentage of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI50 is defined as a ≥ 50% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 41.3 | 64.2 | 70.3
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.47 to 4.49]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.56, 95% CI 2-sided [2.00 to 6.32]

10. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 2.8 | 3.7 | 8.1
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.715, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.32 to 5.31]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.083, Regression, Logistic; Odds Ratio (OR) = 3.02, 95% CI 2-sided [0.86 to 10.56]

11. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 SCORAD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 90 | 100 | 99
units on a scale | -21.40 (1.941) | -29.88 (1.867) | -35.78 (1.862)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -8.48, 95% CI 2-sided [-13.72 to -3.24], Standard Error of Mean 2.663
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -14.38, 95% CI 2-sided [-19.62 to -9.14], Standard Error of Mean 2.662

12. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease: (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD90 is defined as a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 0.9 | 3.7 | 7.2
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.204, Regression, Logistic; Odds Ratio (OR) = 3.21, 95% CI 2-sided [0.53 to 19.37]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.025, Regression, Logistic; Odds Ratio (OR) = 6.99, 95% CI 2-sided [1.27 to 38.53]

13. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: The BSA affected by AD will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage will be reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions. Use the percentage of skin affected for each region (0 to 100%) in EASI as follows: BSA Total = 0.1*BSAhead and neck + 0.3*BSAtrunk + 0.2* BSAupper limbs + 0.4*BSAlower limbs.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 BSA data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 90 | 100 | 100
units on a scale | -18.03 (1.888) | -27.00 (1.825) | -29.73 (1.814)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -8.97, 95% CI 2-sided [-14.07 to -3.87], Standard Error of Mean 2.591
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -11.69, 95% CI 2-sided [-16.78 to -6.61], Standard Error of Mean 2.584

14. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment.
Time Frame: Week 16
Population: All randomized participants who receive at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 108 | 109 | 111
percentage of participants | 2.8 | 4.6 | 2.7
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.721, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p > 0.999, Fisher Exact

15. Secondary Outcome: Mean Gram Quantity of Moderate Potency Background Topical Corticosteroid (TCS) Used (Tube Weights)
Description: Average weights of full tubes were used to determine the dispensed weights for each region. Returned tubes were weighed with cap without carton to determine the amount of TCS in grams (g) used at each visit. Analysis was done via analysis of variance (ANOVA), with geographic region, baseline disease severity (IGA) and treatment as factors in the model.
Time Frame: Week 0 through Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
grams | 252.75 (17.536) | 187.59 (17.508) | 161.61 (17.280)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.0073, ANOVA; Mean Difference (Final Values) = -65.16, 95% CI 2-sided [-112.87 to -17.65], Standard Error of Mean 24.149
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.0002, ANOVA; Mean Difference (Final Values) = -91.14, 95% CI 2-sided [-138.43 to -43.85], Standard Error of Mean 24.038

16. Secondary Outcome: Percent Change From Baseline in Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 98 | 94
percent change | -27.00 (3.370) | -43.44 (3.263) | -51.22 (3.280)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -16.44, 95% CI 2-sided [-25.60 to -7.27], Standard Error of Mean 4.658
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -24.22, 95% CI 2-sided [-33.42 to -15.03], Standard Error of Mean 4.672

17. Secondary Outcome: Change From Baseline in the Total Score of the Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 POEM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 99 | 99
units on a scale | -5.60 (0.764) | -8.50 (0.736) | -10.83 (0.730)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -2.90, 95% CI 2-sided [-4.96 to -0.84], Standard Error of Mean 1.046
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.23, 95% CI 2-sided [-7.28 to -3.18], Standard Error of Mean 1.043

18. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity-Atopic Dermatitis (PGI-S-AD) Score
Description: The PGI-S-AD is a single-item question asking the participant how they would rate their overall AD symptoms over the past 24 hours, using a daily diary. The 5 categories of responses are "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe."
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 PGI-S-AD.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 98 | 94
units on a scale | -0.69 (0.094) | -1.06 (0.091) | -1.18 (0.091)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.63 to -0.12], Standard Error of Mean 0.130
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.75 to -0.24], Standard Error of Mean 0.130

19. Secondary Outcome: Change From Baseline on the Hospital Anxiety Depression Scale (HADS)
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 item questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants Week 16 HADS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 88 | 99 | 99
units on a scale
  Depression | -1.31 (0.311) | -2.05 (0.298) | -2.33 (0.296)
  Anxiety | -1.89 (0.304) | -2.70 (0.292) | -2.80 (0.289)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.083, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.57 to 0.10], Standard Error of Mean 0.425
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.85 to -0.19], Standard Error of Mean 0.423
Statistical Analysis 3: Comparison: Placebo vs 2 mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.63 to 0.00], Standard Error of Mean 0.415
Statistical Analysis 4: Comparison: Placebo vs 4 mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.028, Mixed Models Analysis; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.72 to -0.10], Standard Error of Mean 0.413

20. Secondary Outcome: Change From Baseline on the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, participant-administered,10 question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and at unanswered ("not relevant") responses scored as "0." Scores range from 0 to 30 (less to more impairment), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 DLQI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 99 | 99
units on a scale | -5.58 (0.608) | -7.50 (0.584) | -8.89 (0.851)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-3.56 to -0.28], Standard Error of Mean 0.832
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-4.94 to -1.68], Standard Error of Mean 0.829

21. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) Questionnaire
Description: The WPAI-AD participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 WPAI-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 87 | 99 | 98
units on a scale
  Absenteeism: number analyzed (Participants) | 47 | 57 | 57
  Absenteeism | -6.27 (1.897) | -4.25 (1.741) | -5.29 (1.737)
  Presenteeism: number analyzed (Participants) | 46 | 54 | 54
  Presenteeism | -13.15 (3.203) | -21.28 (2.978) | -23.89 (2.955)
  Work Productivity Loss: number analyzed (Participants) | 46 | 54 | 54
  Work Productivity Loss | -14.25 (3.300) | -22.17 (3.070) | -24.96 (3.051)
  Activity Impairment | -16.75 (2.570) | -26.55 (2.458) | -27.25 (2.447)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Absenteeism; Test type: Superiority; p = 0.435, Mixed Models Analysis; Mean Difference (Final Values) = 2.01, 95% CI 2-sided [-3.06 to 7.08], Standard Error of Mean 2.569
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Absenteeism; Test type: Superiority; p = 0.706, Mixed Models Analysis; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-4.10 to 6.04], Standard Error of Mean 2.569
Statistical Analysis 3: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority — Presenteeism; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = -8.12, 95% CI 2-sided [-16.78 to 0.54], Standard Error of Mean 4.384
Statistical Analysis 4: Comparison: Placebo vs 4 mg Baricitinib; Presenteeism; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = -10.73, 95% CI 2-sided [-19.30 to -2.17], Standard Error of Mean 4.336
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority — Work Productivity Loss; p = 0.081, Mixed Models Analysis; Mean Difference (Final Values) = -7.93, 95% CI 2-sided [-16.84 to 0.99], Standard Error of Mean 4.511
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; Work productivity Loss; Test type: Superiority; p = 0.018, Mixed Models Analysis; Mean Difference (Final Values) = -10.71, 95% CI 2-sided [-19.55 to 1.88], Standard Error of Mean 4.473
Statistical Analysis 7: Comparison: Placebo vs 2 mg Baricitinib; Activity Impairment; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -9.80, 95% CI 2-sided [-16.71 to -2.89], Standard Error of Mean 3.511
Statistical Analysis 8: Comparison: Placebo vs 4 mg Baricitinib; Activity Impairment; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -10.50, 95% CI 2-sided [-17.39 to -3.61], Standard Error of Mean 3.500

22. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm
Description: The EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EQ-5D-5L Health State Index US and UK data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 87 | 99 | 98
units on a scale
  Health State Index Score (US Algorithm) | 0.09 (0.013) | 0.12 (0.012) | 0.14 (0.012)
  Health State Index Score (UK Algorithm) | 0.13 (0.018) | 0.17 (0.017) | 0.21 (0.017)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Health State Index US; Test type: Superiority; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.06], Standard Error of Mean 0.017
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Health State Index US; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.02 to 0.09], Standard Error of Mean 0.017
Statistical Analysis 3: Comparison: Placebo vs 2 mg Baricitinib; Health State Index UK; Test type: Superiority; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.08], Standard Error of Mean 0.024
Statistical Analysis 4: Comparison: Placebo vs 4 mg Baricitinib; Health State Index UK; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.02 to 0.12], Standard Error of Mean 0.024

23. Secondary Outcome: Change From Baseline on the EQ-5D-5L Visual Analog Scale (VAS)
Description: The EQ-5D-5L is a 2-part measurement. The second part is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EQ-5D-5L VAS data.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 87 | 99 | 98
millimeters | 11.00 (1.903) | 15.12 (1.806) | 17.06 (1.805)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.113, Mixed Models Analysis; Mean Difference (Final Values) = 4.12, 95% CI 2-sided [-0.98 to 9.23], Standard Error of Mean 2.593
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = 6.06, 95% CI 2-sided [0.96 to 11.16], Standard Error of Mean 2.592

24. Secondary Outcome: Mean Number of Days Without Use of Background TCS
Description: The ANCOVA model includes treatment, region, and baseline disease severity (IGA) as factors.
Time Frame: Week 0 through Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
days | 12.45 (3.17) | 22.49 (3.16) | 29.78 (3.12)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.022, ANCOVA; Mean Difference (Final Values) = 10.04, 95% CI 2-sided [1.46 to 18.36], Standard Error of Mean 4.36
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 17.33, 95% CI 2-sided [8.79 to 25.88], Standard Error of Mean 4.34

25. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a ≥ 2 Point Improvement
Description: as for outcome 10
Time Frame: Week 4
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 109 | 109 | 111
percentage of participants | 5.5 | 17.4 | 19.8
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 3.83, 95% CI 2-sided [1.46 to 10.03]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [1.77 to 11.87]

ADVERSE EVENTS:
Time Frame: Baseline up to 20 weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/109 | 0/111
Serious Adverse Events (participants affected / at risk) | 4/108 | 2/109 | 4/111
Other Adverse Events (participants affected / at risk) | 15/108 | 24/109 | 26/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | 2 mg Baricitinib (N=109) | 4 mg Baricitinib (N=111)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye infection toxoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | 2 mg Baricitinib (N=109) | 4 mg Baricitinib (N=111)
Folliculitis (Infections and infestations) | 0 (0) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 13 (14) | 12 (16) | 17 (18)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 8 (12) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT03733301/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03733301/SAP_001.pdf